CLINICAL TRIAL: NCT01841203
Title: Evaluation of a Rapid Dual Point-of-care Assay for Targeting Antibiotic Treatment for Yaws Eradication: a Prospective Descriptive Study
Brief Title: Dual Point-of-care Test for the Diagnosis of Yaws
Acronym: YARADI
Status: Completed | Type: Observational
Sponsor: Oriol Mitja (Other)
Collaborators: Papua New Guinea Institute of Medical Research (Other Government); Papua New Guinea National Department of Health, Disease Control (Unknown); Divine Word University (Unknown); Barcelona Centre for International Health Research (Other)
Responsible Party: Sponsor-Investigator, Oriol Mitja, MD, Lihir Medical Centre
Organization: Lihir Medical Centre (Other)
Other Study IDs: YARADI
Record Dates: First submitted 2013-04-19; First posted 2013-04-26 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Yaws
Keywords: Diagnosis; Rapid tests; non-treponemal serology; eradication
MeSH Terms: conditions — Yaws; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DPP/RPR-TPHA comparison: The evaluation of T1 (treponemal line) will be conducted by using the T1 positivity identified by naked eye or automated reader to compare with that of TPHA; while the evaluation of T2 (non-treponemal line) will be conducted by using the T2 positivity identified by naked eye, or automatic reader at cut-off value of 20, to compare with the result of RPR.

SUMMARY:
A dual POC immunoassay simultaneously detecting non-treponemal and treponemal antibodies was developed for the diagnosis of infections with T. pallidum. The assay is designed for use in resource-limited settings where challenging conditions (such as lack of electricity, running water, or laboratory equipment) commonly exist. We sought to compare performance of the dual-POC assay for diagnosis of yaws infection with that of the RPR and TPHA as reference standards.

DETAILED DESCRIPTION:
Yaws is an infectious disease caused by Treponema pallidum subspecies pertenue, a bacterium which closely resembles the causative agent of syphilis, and is spread by skin to skin contact. In the field, yaws is diagnosed on the basis of epidemiological context, evocative symptoms and signs and positive serological tests or dark field microscopy. The darkfield microscopy is not easy to perform , hence the interest in serological tests. The serological tests used to confirm yaws are the same as those used to diagnose syphilis. Yaws serologic diagnosis relies on testing for non-treponemal and treponemal antibodies. These antibodies differ markedly with respect to antigenic reactivities and kinetics during the disease process.

Historically screening for yaws has involved the use of nontreponemal tests, such as rapid plasma reagin or venereal disease research laboratory. Positive results of nontreponemal tests of specimens are then confirmed using a more specific treponemal test, such as Treponema pallidum haemagglutination. However, the equipment and personnel requirements for conducting and interpreting these laboratory-tests are rarely available in low-resource settings in developing countries where yaws occurs.

Rapid treponemal tests which detect antibodies to T. pallidum antigen have become popular for the diagnosis of venereal syphilis due to their many advantages. These tests that can be performed outside a laboratory setting with minimal training and using blood collected by a finger prick, which makes them extremely useful in remote areas where laboratories are not available. However, the rapid treponemal tests for syphilis detect treponemal antibodies, which limits their use for interpretation of the disease status since they cannot distinguish between active and past or treated infection.

A combined point-of-care (POC) test which detects both treponemal and non-treponemal antibodies has recently been evaluated for the diagnosis of syphilis, and appears promising for yaws diagnosis. The use of the dual POC test would result in the ability to both screen and confirm the serological status of patients with suspected yaws within 15 minutes and give a better indication of active disease.

ELIGIBILITY:
Inclusion Criteria:

* Children from 2 to 15 years with clinical suspicion of active yaws

Exclusion Criteria:

* Persons who are unable to sustain venipuncture; persons who do not provide an informed consent, or withdraw consent

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients will be recruited from Lihir Island villages in April 2013. This community has been described previously. We will conduct community-based surveys and we invited children aged 1 - 15 years suspected to have yaws by clinical examination to participate in the study. All children for whom a parent or guardian gives written informed consent will be included consecutively
Sampling Method: Non-Probability Sample
Enrollment: 703 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To determine the accuracy of the dual-test as compared to recognized standard methods | 1 month
  Sensitivity and Specificity as compared to RPR and TPHA
  1. Proportion of actual TPHA/RPR positives which are correctly identified as such by DPP (dual-test)T1 and T2 respectively
  2. Proportion of TPHA/RPR negatives which are correctly identified as such by DPP (dual-test)T1 and T2 respectively

SECONDARY OUTCOMES:
Accuracy of DPP in whole blood and plasma | 1 month
  Specimens will be randomly tested using DPP, either in plasma or blood.
  Sensitivity and Specificity of DPP in whole blood and DPP in plasma will be compared.
Accuracy of DPP determined by Naked eye and Reader | 1 month
  Specimens will be tested using DPP, read by naked eye and also using automated reader.
  Sensitivity and Specificity of DPP result read by naked eye and DPP using automated reader will be compared.

CONTACTS AND LOCATIONS:
Locations (2):
- Papua New Guinea (2):
  - Karkar Island, Marup Village, Madang Province
  - Lihir Medical Centre, Londolovit, New Ireland Province

REFERENCES:
- [Derived] Ayove T, Houniei W, Wangnapi R, Bieb SV, Kazadi W, Luke LN, Manineng C, Moses P, Paru R, Esfandiari J, Alonso PL, de Lazzari E, Bassat Q, Mabey D, Mitja O. Sensitivity and specificity of a rapid point-of-care test for active yaws: a comparative study. Lancet Glob Health. 2014 Jul;2(7):e415-21. doi: 10.1016/S2214-109X(14)70231-1. Epub 2014 May 31. PMID 25103395